CLINICAL TRIAL: NCT07224659
Title: Exercise and Mortality in Middle-Aged and Older Adults: A Target Trial Emulation
Brief Title: Exercise and Mortality in Middle-Aged and Older Adults
Status: Not yet recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 25603
Record Dates: First submitted 2025-11-02; First posted 2025-11-05 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Overall Survival (All-cause Mortality)
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1 - Control: 0 or less than 1 day per week, with each session, on average < 15 minutes.
  Interventions: Behavioral: Control
- Arm 2 - Exercise: >/= 2 days per week of moderate or vigorous intensity, with each session, on average, >/=20 minutes in duration.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Control — 0 or less than 1 day per week, with each session, on average < 15 minutes.
  Groups: Arm 1 - Control
Behavioral: Exercise — >/= 2 days per week of moderate or vigorous intensity, with each session, on average, >/=20 minutes in duration.
  Groups: Arm 2 - Exercise

SUMMARY:
This protocol is a retrospective study using the observational data of the the Prostate, Lung, Colorectal, and Ovarian (PLCO) screening trial with over 150,000 participants aged 55-74 years to conduct a target trial emulation to examine the association between self-reported exercise and all cause and cause-specific mortality in apparently healthy, middle-aged and older adults. The PLCO includes assessments of participants' exercise level at two timepoints: at randomization into the PLCO trial (Q0) and 5-7 years after randomization into the PLCO (Q1).

ELIGIBILITY:
* Adults enrolled into the PLCO screening trial.
* Among participants reporting low exercise at Q0 (i.e., 0 or less than 1 day/week, with each session <15 minutes in duration), completion of an exercise survey at Q1 as part of PLCO standard trial procedures no later than 5 years after reporting non-exercising status [i.e., no exercise) at Q0.
* No evidence of any of the following absolute contraindications to exercise: uncontrolled hypertension, symptomatic valvular disease; hypertrophic cardiomyopathy; unstable angina pectoris; primary pulmonary hypertension; heart failure; severe arrhythmia; diagnosed dementia; any form of cancer other than non-melanoma, and severe infectious disease.

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults enrolled into the PLCO screening trial
Sampling Method: Non-Probability Sample
Enrollment: 19000 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-08-06 (Estimated); Study Completion 2026-08-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival (all-cause mortality) | up to 19 years
  All-cause mortality (death from any cause) occurring within the follow-up period in the PLCO screening trial.
Cause-specific mortality | up to 19 years
  Cause-specific mortality (cancer mortality, mortality from other causes) occurring within the total follow-up period in the PLCO screening trial.

SECONDARY OUTCOMES:
Cancer incidence | up to 19 years
  Cancer incidence occurring within the total follow-up period in the PLCO screening trial.

OTHER OUTCOMES:
Exploratory Analyses #1 | up to 19 years
  Analyses to examine whether the association between exercise vs. control with all-cause mortality differs as a function of:
  * Sex (male vs. female)
  * Age (<50 years vs. =/>50 years)
Exploratory Analyses #2 | up to 19 years
  Examine the association between exercise vs. control with incidence of individual cancer types.

CONTACTS AND LOCATIONS:
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: Undecided